CLINICAL TRIAL: NCT04165473
Title: A Training Program for Developing Social- and Personal Resources and Its Effects on Emotional, Physical and Social Wellbeing in Adults
Brief Title: A Training Program for Developing Social- and Personal Resources
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christoph Janka, Principal Investigator, Medical University of Vienna
Other Study IDs: EK1592/2019
Record Dates: First submitted 2019-11-08; First posted 2019-11-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Stress, Psychological; Stress, Emotional; Health Behavior; Satisfaction, Personal; Somatic Symptom; Psychophysiology; Family Relations; Program Evaluation
Keywords: Training Program; Personal Resources; Social Resources; Adults; Emotional Wellbeing; Physical Wellbeing; Social Wellbeing; Perceived Stress; Satisfaction with Life; Health Behavior; Quality of Relationships; Somatic Symptoms; Sense of Coherence; Life Goals; Meaning in Life; Transcendence; Evaluation
MeSH Terms: conditions — Stress, Psychological; Health Behavior; Personal Satisfaction; Medically Unexplained Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Study participants having finished the following course in the past will be assigned to the intervention group: During a 6-module course, with four 3-day modules and two 5-day modules in the timeframe of one year, participants learn ways to strengthen their personal resources to establish effective social relationships and to develop skills as a social being. In between the module courses, the participants take 5 single sessions with an instructed trainer and document 10 conversations/social situations where they successfully applied the new skills.
  Interventions: Behavioral: Training Program for Developing Social- and Personal Resources
- Control Group: Individuals without intervention

INTERVENTIONS:
Behavioral: Training Program for Developing Social- and Personal Resources — The training-method shows how one's own resonance can be exposed in order to live the balance between one's own needs and those of others.
  Living one's own resonance means: more quality of life, work-life balance, holistic health through living feelings and talents, live equal, respectful and loving relationships, more personal responsibility, authentic decision making find new role models in private and professional areas.
  The teaching and learning methods of the trainings and seminars are implemented according to the latest state of brain research and enable new perspectives with regard to new learning strategies, goals, enthusiasm and motivation.
  With the Kutschera-Resonanz® method we teach and learn to consciously use this unconscious reservoir so that completely new dimensions in thinking and acting open up.
  In this training program the basic tools of communication and interaction according to the Kutschera-Resonanz® method are taught and experienced by the participants.
  Other Names: Kutschera-Resonance-Practitioner
  Groups: Intervention Group

SUMMARY:
In this study, a new psychosocial training for social relationships for adults will be evaluated. In a 6-module course, with four 3-day modules and two 5-day modules in the timeframe of one year, participants learn ways to strengthen their personal resources to establish effective social relationships and to develop skills as a social being. In between the module courses, the participants take 5 single sessions with an instructed trainer and document 10 conversations/social situations where they successfully apply the acquired personal and social skills. For my study, I will recruit a total of 200 persons. Approx. one hundred participants for the intervention group and 100 individuals for the control group. During the course of the training, the participants are taught social and personal skills that should result in a lower perceived stress level in daily life, improved health behaviour, a decreased presence of common somatic symptoms, a higher satisfaction with their lives, improved quality of their social relationships and a higher wellbeing. Data from study participants having accomplished additional training programs with the same training provider will be used to evaluate the influence on the results compared to participants without the extra addition for this study.

The training participants will be assessed together with the controls. All study participants will be evaluated with standardized online questionnaires.

DETAILED DESCRIPTION:
Human beings perceive stress differently and several bio-psycho-social factors, as well as personal and environmental factors influence how persons can manage and cope with stress. Concepts, such as resilience, facilitate positive attitudes towards self-management of stressful life situations. Phylogenetically, (positive) stress produced/s adequate reactions of humans in difficult or dangerous situations, like to fight or run away in the time when human beings were predominantly hunter-gatherers. However, persistent stress, as well as the inability to sufficiently cope with stress have several negative consequences for the physical and mental health of humans. Negative stress is a major contributor to chronic diseases, like cardiovascular diseases, cancer, respiratory disorders, mental diseases including depression, but also the occurrence of accidental injuries. Insufficient coping can result in a harmful health behaviour at first and in the long term to a higher overall morbidity and mortality. This means not only a personal, emotional and physical burden but also a financial burden for the society as a whole, as well as the health system of a country.

On the other hand, satisfactory social relationships were found to have a stress buffering, positive effect on how people deal with stress and are beneficial for one's own health over the course of life. Satisfactory social relationships might even lead to longevity.

The following research questions will be addressed in this study:

1. What effect has a 1-year training program for social- and personal resources A) on the outcome parameters perceived stress level, health behavior, presence of common somatic symptoms, satisfaction with life, quality of social relationships, wellbeing compared to a control group? B) on the perception of the trainings aims life goals, meaning in life, sense of coherence, social- and personal resources and transcendence of the participants compared to a control group? C) and how do sociodemographic characteristics influence these effects?
2. If changes occur A) what effect has the time passed since finishing the training on the outcome parameters and training aims in participants? B) what effect has the time passed since finishing the training on the outcome parameters and aims in participants compared to the control group?
3. How are the perceptions of the training aims (concerning life goals, meaning in life, sense of coherence, social- and personal resources and transcendence) related to perceived stress level, health behaviour, health status, satisfaction with life, quality of social relationships, and wellbeing and how much does each of them contribute?
4. What effect has the exposure to this training content (number of trainings and seminars taken) on the outcome parameters and training aims A) in training participants? B) compared to the control group?
5. What kind of statistically relevant effects are present for the combination and interaction of the training aims and sociodemographic characteristics on the outcome variables?

ELIGIBILITY:
Inclusion Criteria:

* male, female, other
* fluently German speaking
* between 18-70 years of age
* given informed consent

Intervention Arm:

- having completed the "Resonanz Practitioner" training

Exclusion Criteria:

- taking too long or too little time to finish the questionnaire (> 3 standard deviations)

* wrong answer on the control question
* where no time stamp available, check for suspicious patterns and drop-out if they are present

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals from the general population with the intervention group having finished the "Resonanz Practitioner" training at Institut Kutschera.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Level | Assessed on Day 1
  "Perceived Stress Scale" score (PSS) difference between Intervention and Control Group, score range 0-40 where a lower score means less perceived stress

SECONDARY OUTCOMES:
Health behavior | Assessed on Day 1
  Difference in "Fragebogen zur Erfassung des Gesundheitsverhaltens" (FEG) scores for health behavior between intervention and control group, score range: sleep: 10-50, physical activity: -20-26, psychosocial burden: 2-46, where higher scores mean more positive behavior
Presence of common somatic symptoms | Assessed on Day 1
  Difference in "Fragebogen zur Erfassung des Gesundheitsverhaltens" (FEG) scores for Presence of common somatic symptoms between intervention and control group, score range: 5-25, where a lower score means less symptoms
Wellbeing | Assessed on Day 1
  Difference in scores for Wellbeing (WHO-5) between intervention and control group, score range: 0-25, with higher scores meaning better wellbeing
Quality of Relationships | Assessed on Day 1
  Difference in scores for Quality of Relationships - Evaluation of Social Systems Scale (EVOS) and Experience in Social Systems Scale (EXIS) between intervention and control group, EVOS score range: 0-3, EXIS score range: 1-6, with higher scores meaning better Quality of Relationships
Satisfaction with Life | Assessed on Day 1
  Difference in Life Satisfaction Scale (LS-4) scores between intervention and control group, score range: 4-20 with higher scores meaning better satisfaction with life

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Janka, DI, Principal Investigator — Medical Universtiy of Vienna
Locations (1):
- Medical Universtiy of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen S, Wills TA. Stress, social support, and the buffering hypothesis. Psychol Bull. 1985 Sep;98(2):310-57. No abstract available. PMID 3901065
- [Background] House JS, Landis KR, Umberson D. Social relationships and health. Science. 1988 Jul 29;241(4865):540-5. doi: 10.1126/science.3399889.
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] Sebanz N, Bekkering H, Knoblich G. Joint action: bodies and minds moving together. Trends Cogn Sci. 2006 Feb;10(2):70-6. doi: 10.1016/j.tics.2005.12.009. Epub 2006 Jan 10. PMID 16406326
- [Background] Garrod S, Pickering MJ. Joint action, interactive alignment, and dialog. Top Cogn Sci. 2009 Apr;1(2):292-304. doi: 10.1111/j.1756-8765.2009.01020.x. PMID 25164934
- [Background] Melis AP. The evolutionary roots of human collaboration: coordination and sharing of resources. Ann N Y Acad Sci. 2013 Sep;1299:68-76. doi: 10.1111/nyas.12263. PMID 25708081
- [Background] Melis AP, Grocke P, Kalbitz J, Tomasello M. One for You, One for Me: Humans' Unique Turn-Taking Skills. Psychol Sci. 2016 Jul;27(7):987-96. doi: 10.1177/0956797616644070. Epub 2016 May 25. PMID 27225221
- [Background] Melis AP, Semmann D. How is human cooperation different? Philos Trans R Soc Lond B Biol Sci. 2010 Sep 12;365(1553):2663-74. doi: 10.1098/rstb.2010.0157. PMID 20679110
- [Background] Warneken F, Tomasello M. Altruistic helping in human infants and young chimpanzees. Science. 2006 Mar 3;311(5765):1301-3. doi: 10.1126/science.1121448. PMID 16513986
- [Background] Warneken F, Tomasello M. The roots of human altruism. Br J Psychol. 2009 Aug;100(Pt 3):455-71. doi: 10.1348/000712608X379061. Epub 2008 Dec 5. PMID 19063815
- [Background] Nelson SK, Layous K, Cole SW, Lyubomirsky S. Do unto others or treat yourself? The effects of prosocial and self-focused behavior on psychological flourishing. Emotion. 2016 Sep;16(6):850-61. doi: 10.1037/emo0000178. Epub 2016 Apr 21. PMID 27100366
- [Background] Wedekind C, Braithwaite VA. The long-term benefits of human generosity in indirect reciprocity. Curr Biol. 2002 Jun 25;12(12):1012-5. doi: 10.1016/s0960-9822(02)00890-4. PMID 12123575
- [Background] Scott S, Knapp M, Henderson J, Maughan B. Financial cost of social exclusion: follow up study of antisocial children into adulthood. BMJ. 2001 Jul 28;323(7306):191. doi: 10.1136/bmj.323.7306.191. PMID 11473907
- [Background] Cacioppo JT, Hawkley LC, Crawford LE, Ernst JM, Burleson MH, Kowalewski RB, Malarkey WB, Van Cauter E, Berntson GG. Loneliness and health: potential mechanisms. Psychosom Med. 2002 May-Jun;64(3):407-17. doi: 10.1097/00006842-200205000-00005. PMID 12021415
- [Background] Paradis AD, Koenen KC, Fitzmaurice GM, Buka SL. Impact of persistent and adolescent-limited antisocial behaviour on adult health outcomes. J Epidemiol Community Health. 2016 Oct;70(10):1004-10. doi: 10.1136/jech-2014-205140. Epub 2016 Apr 11. PMID 27069087
- [Background] Twenge JM, Baumeister RF, DeWall CN, Ciarocco NJ, Bartels JM. Social exclusion decreases prosocial behavior. J Pers Soc Psychol. 2007 Jan;92(1):56-66. doi: 10.1037/0022-3514.92.1.56. PMID 17201542
- [Background] Layous K, Chancellor J, Lyubomirsky S. Positive activities as protective factors against mental health conditions. J Abnorm Psychol. 2014 Feb;123(1):3-12. doi: 10.1037/a0034709. PMID 24661154
- [Background] Uchino BN. Social support and health: a review of physiological processes potentially underlying links to disease outcomes. J Behav Med. 2006 Aug;29(4):377-87. doi: 10.1007/s10865-006-9056-5. Epub 2006 Jun 7. PMID 16758315
- [Background] Ackard DM, Neumark-Sztainer D, Story M, Perry C. Parent-child connectedness and behavioral and emotional health among adolescents. Am J Prev Med. 2006 Jan;30(1):59-66. doi: 10.1016/j.amepre.2005.09.013. PMID 16414425
- [Background] Procidano ME, Heller K. Measures of perceived social support from friends and from family: three validation studies. Am J Community Psychol. 1983 Feb;11(1):1-24. doi: 10.1007/BF00898416. PMID 6837532
- [Background] Ren XS. Marital status and quality of relationships: the impact on health perception. Soc Sci Med. 1997 Jan;44(2):241-9. doi: 10.1016/s0277-9536(96)00158-x. PMID 9015876
- [Background] Gouin JP, Carter CS, Pournajafi-Nazarloo H, Glaser R, Malarkey WB, Loving TJ, Stowell J, Kiecolt-Glaser JK. Marital behavior, oxytocin, vasopressin, and wound healing. Psychoneuroendocrinology. 2010 Aug;35(7):1082-90. doi: 10.1016/j.psyneuen.2010.01.009. Epub 2010 Feb 9. PMID 20144509
- [Background] Kiecolt-Glaser JK, Gouin JP, Hantsoo L. Close relationships, inflammation, and health. Neurosci Biobehav Rev. 2010 Sep;35(1):33-8. doi: 10.1016/j.neubiorev.2009.09.003. Epub 2009 Sep 12. PMID 19751761
- [Background] Kiecolt-Glaser JK, McGuire L, Robles TF, Glaser R. Emotions, morbidity, and mortality: new perspectives from psychoneuroimmunology. Annu Rev Psychol. 2002;53:83-107. doi: 10.1146/annurev.psych.53.100901.135217. PMID 11752480
- [Background] Seeman TE. Social ties and health: the benefits of social integration. Ann Epidemiol. 1996 Sep;6(5):442-51. doi: 10.1016/s1047-2797(96)00095-6. PMID 8915476
- [Background] Waldinger RJ, Cohen S, Schulz MS, Crowell JA. Security of attachment to spouses in late life: Concurrent and prospective links with cognitive and emotional wellbeing. Clin Psychol Sci. 2015 Jun 1;3(4):516-529. doi: 10.1177/2167702614541261. PMID 26413428
- [Background] Chopik WJ, O'Brien E. Happy you, healthy me? Having a happy partner is independently associated with better health in oneself. Health Psychol. 2017 Jan;36(1):21-30. doi: 10.1037/hea0000432. Epub 2016 Sep 19. PMID 27642761
- [Background] Roberson PNE, Shorter RL, Woods S, Priest J. How health behaviors link romantic relationship dysfunction and physical health across 20 years for middle-aged and older adults. Soc Sci Med. 2018 Mar;201:18-26. doi: 10.1016/j.socscimed.2018.01.037. Epub 2018 Feb 3. PMID 29427892
- [Background] Rydstedt LW, Head J, Stansfeld SA, Woodley-Jones D. Quality of workplace social relationships and perceived health. Psychol Rep. 2012 Jun;110(3):781-90. doi: 10.2466/01.13.21.PR0.110.3.781-790. PMID 22897084
- [Background] Uchino BN, Cawthon RM, Smith TW, Light KC, McKenzie J, Carlisle M, Gunn H, Birmingham W, Bowen K. Social relationships and health: is feeling positive, negative, or both (ambivalent) about your social ties related to telomeres? Health Psychol. 2012 Nov;31(6):789-96. doi: 10.1037/a0026836. Epub 2012 Jan 9. PMID 22229928
- [Background] Fredrickson BL. The role of positive emotions in positive psychology. The broaden-and-build theory of positive emotions. Am Psychol. 2001 Mar;56(3):218-26. doi: 10.1037//0003-066x.56.3.218. PMID 11315248
- [Background] Pressman SD, Cohen S. Does positive affect influence health? Psychol Bull. 2005 Nov;131(6):925-971. doi: 10.1037/0033-2909.131.6.925. PMID 16351329
- [Background] Wang CS, Kenneth T, Ku G, Galinsky AD. Perspective-taking increases willingness to engage in intergroup contact. PLoS One. 2014 Jan 22;9(1):e85681. doi: 10.1371/journal.pone.0085681. eCollection 2014. PMID 24465648
- [Background] Ruiz-Aranda D, Extremera N, Pineda-Galan C. Emotional intelligence, life satisfaction and subjective happiness in female student health professionals: the mediating effect of perceived stress. J Psychiatr Ment Health Nurs. 2014 Mar;21(2):106-13. doi: 10.1111/jpm.12052. Epub 2013 Apr 12. PMID 23578272
- [Background] Yang SX, Jowett S, Chan DK. Effects of big-five personality traits on the quality of relationship and satisfaction in Chinese coach-athlete dyads. Scand J Med Sci Sports. 2015 Aug;25(4):568-80. doi: 10.1111/sms.12329. Epub 2014 Nov 4. PMID 25367655
- [Background] Gudsnuk K, Champagne FA. Epigenetic influence of stress and the social environment. ILAR J. 2012;53(3-4):279-88. doi: 10.1093/ilar.53.3-4.279. PMID 23744967
- [Background] Daskalakis NP, Bagot RC, Parker KJ, Vinkers CH, de Kloet ER. The three-hit concept of vulnerability and resilience: toward understanding adaptation to early-life adversity outcome. Psychoneuroendocrinology. 2013 Sep;38(9):1858-73. doi: 10.1016/j.psyneuen.2013.06.008. Epub 2013 Jul 7. PMID 23838101
- [Background] Romeo RD. Perspectives on stress resilience and adolescent neurobehavioral function. Neurobiol Stress. 2014 Nov 8;1:128-33. doi: 10.1016/j.ynstr.2014.11.001. eCollection 2015 Jan. PMID 27589663
- [Background] Masten AS. Ordinary magic. Resilience processes in development. Am Psychol. 2001 Mar;56(3):227-38. doi: 10.1037//0003-066x.56.3.227. PMID 11315249
- [Background] Kobasa SC. Stressful life events, personality, and health: an inquiry into hardiness. J Pers Soc Psychol. 1979 Jan;37(1):1-11. doi: 10.1037//0022-3514.37.1.1. PMID 458548
- [Background] Baram TZ, Davis EP, Obenaus A, Sandman CA, Small SL, Solodkin A, Stern H. Fragmentation and unpredictability of early-life experience in mental disorders. Am J Psychiatry. 2012 Sep;169(9):907-15. doi: 10.1176/appi.ajp.2012.11091347. PMID 22885631
- [Background] Krugers HJ, Arp JM, Xiong H, Kanatsou S, Lesuis SL, Korosi A, Joels M, Lucassen PJ. Early life adversity: Lasting consequences for emotional learning. Neurobiol Stress. 2016 Nov 27;6:14-21. doi: 10.1016/j.ynstr.2016.11.005. eCollection 2017 Feb. PMID 28229105
- [Background] Seedat S, Stein DJ, Jackson PB, Heeringa SG, Williams DR, Myer L. Life stress and mental disorders in the South African stress and health study. S Afr Med J. 2009 May;99(5 Pt 2):375-82. PMID 19588801
- [Background] Ansell EB, Gu P, Tuit K, Sinha R. Effects of cumulative stress and impulsivity on smoking status. Hum Psychopharmacol. 2012 Mar;27(2):200-8. doi: 10.1002/hup.1269. PMID 22389084
- [Background] Laloyaux J, Dessart G, Van der Linden M, Lemaire M, Laroi F. Maladaptive emotion regulation strategies and stress sensitivity mediate the relation between adverse life events and attenuated positive psychotic symptoms. Cogn Neuropsychiatry. 2016;21(2):116-29. doi: 10.1080/13546805.2015.1137213. Epub 2016 Feb 1. PMID 26829655
- [Background] Woodhead EL, Cronkite RC, Moos RH, Timko C. Coping strategies predictive of adverse outcomes among community adults. J Clin Psychol. 2014 Dec;70(12):1183-95. doi: 10.1002/jclp.21924. Epub 2013 Apr 29. PMID 23629952
- [Background] Littleton H, Horsley S, John S, Nelson DV. Trauma coping strategies and psychological distress: A meta-analysis. J Trauma Stress. 2007 Dec;20(6):977-88. doi: 10.1002/jts.20276. PMID 18157893
- [Background] Hanssen LM, Schutte NS, Malouff JM, Epel ES. The Relationship Between Childhood Psychosocial Stressor Level and Telomere Length: A Meta-Analysis. Health Psychol Res. 2017 May 16;5(1):6378. doi: 10.4081/hpr.2017.6378. eCollection 2017 May 16. PMID 28603779
- [Background] Schaakxs R, Wielaard I, Verhoeven JE, Beekman AT, Penninx BW, Comijs HC. Early and recent psychosocial stress and telomere length in older adults. Int Psychogeriatr. 2016 Mar;28(3):405-13. doi: 10.1017/S1041610215001155. Epub 2015 Aug 12. PMID 26265356
- [Background] Wu G, Feder A, Cohen H, Kim JJ, Calderon S, Charney DS, Mathe AA. Understanding resilience. Front Behav Neurosci. 2013 Feb 15;7:10. doi: 10.3389/fnbeh.2013.00010. eCollection 2013. PMID 23422934
- [Background] Oliveira BS, Zunzunegui MV, Quinlan J, Fahmi H, Tu MT, Guerra RO. Systematic review of the association between chronic social stress and telomere length: A life course perspective. Ageing Res Rev. 2016 Mar;26:37-52. doi: 10.1016/j.arr.2015.12.006. Epub 2015 Dec 28. PMID 26732034
- [Background] Epel ES, Blackburn EH, Lin J, Dhabhar FS, Adler NE, Morrow JD, Cawthon RM. Accelerated telomere shortening in response to life stress. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17312-5. doi: 10.1073/pnas.0407162101. Epub 2004 Dec 1. PMID 15574496
- [Background] Cohen S, Tyrrell DA, Smith AP. Negative life events, perceived stress, negative affect, and susceptibility to the common cold. J Pers Soc Psychol. 1993 Jan;64(1):131-40. doi: 10.1037//0022-3514.64.1.131. PMID 8421249
- [Background] Buysse DJ. Sleep health: can we define it? Does it matter? Sleep. 2014 Jan 1;37(1):9-17. doi: 10.5665/sleep.3298. PMID 24470692
- [Background] Prather AA, Puterman E, Lin J, O'Donovan A, Krauss J, Tomiyama AJ, Epel ES, Blackburn EH. Shorter leukocyte telomere length in midlife women with poor sleep quality. J Aging Res. 2011;2011:721390. doi: 10.4061/2011/721390. Epub 2011 Oct 20. PMID 22046530
- [Background] Hirotsu C, Tufik S, Andersen ML. Interactions between sleep, stress, and metabolism: From physiological to pathological conditions. Sleep Sci. 2015 Nov;8(3):143-52. doi: 10.1016/j.slsci.2015.09.002. Epub 2015 Sep 28. PMID 26779321
- [Background] Kent RG, Uchino BN, Cribbet MR, Bowen K, Smith TW. Social Relationships and Sleep Quality. Ann Behav Med. 2015 Dec;49(6):912-7. doi: 10.1007/s12160-015-9711-6. PMID 25976874
- [Background] Masoudnia E. Impact of weak social ties and networks on poor sleep quality: A case study of Iranian employees. Asian J Psychiatr. 2015 Dec;18:42-8. doi: 10.1016/j.ajp.2015.10.005. Epub 2015 Oct 19. PMID 26494526
- [Background] Hintsanen M, Puttonen S, Smith K, Tornroos M, Jokela M, Pulkki-Raback L, Hintsa T, Merjonen P, Dwyer T, Raitakari OT, Venn A, Keltikangas-Jarvinen L. Five-factor personality traits and sleep: evidence from two population-based cohort studies. Health Psychol. 2014 Oct;33(10):1214-23. doi: 10.1037/hea0000105. Epub 2014 Aug 18. PMID 25133841
- [Background] Zhi TF, Sun XM, Li SJ, Wang QS, Cai J, Li LZ, Li YX, Xu MJ, Wang Y, Chu XF, Wang ZD, Jiang XY. Associations of sleep duration and sleep quality with life satisfaction in elderly Chinese: The mediating role of depression. Arch Gerontol Geriatr. 2016 Jul-Aug;65:211-7. doi: 10.1016/j.archger.2016.03.023. Epub 2016 Mar 30. PMID 27100684
- [Background] Ben Simon E, Walker MP. Sleep loss causes social withdrawal and loneliness. Nat Commun. 2018 Aug 14;9(1):3146. doi: 10.1038/s41467-018-05377-0. PMID 30108218
- [Background] Puterman E, Lin J, Blackburn E, O'Donovan A, Adler N, Epel E. The power of exercise: buffering the effect of chronic stress on telomere length. PLoS One. 2010 May 26;5(5):e10837. doi: 10.1371/journal.pone.0010837. PMID 20520771
- [Background] Iwasaki Y, Zuzanek J, Mannell RC. The effects of physically active leisure on stress-health relationships. Can J Public Health. 2001 May-Jun;92(3):214-8. doi: 10.1007/BF03404309. PMID 11496634
- [Background] Almeida OP, Khan KM, Hankey GJ, Yeap BB, Golledge J, Flicker L. 150 minutes of vigorous physical activity per week predicts survival and successful ageing: a population-based 11-year longitudinal study of 12 201 older Australian men. Br J Sports Med. 2014 Feb;48(3):220-5. doi: 10.1136/bjsports-2013-092814. Epub 2013 Sep 3. PMID 24002240
- [Background] Arem H, Moore SC, Patel A, Hartge P, Berrington de Gonzalez A, Visvanathan K, Campbell PT, Freedman M, Weiderpass E, Adami HO, Linet MS, Lee IM, Matthews CE. Leisure time physical activity and mortality: a detailed pooled analysis of the dose-response relationship. JAMA Intern Med. 2015 Jun;175(6):959-67. doi: 10.1001/jamainternmed.2015.0533. PMID 25844730
- [Background] Ekblom-Bak E, Ekblom B, Vikstrom M, de Faire U, Hellenius ML. The importance of non-exercise physical activity for cardiovascular health and longevity. Br J Sports Med. 2014 Feb;48(3):233-8. doi: 10.1136/bjsports-2012-092038. Epub 2013 Oct 28. PMID 24167194
- [Background] Bize R, Johnson JA, Plotnikoff RC. Physical activity level and health-related quality of life in the general adult population: a systematic review. Prev Med. 2007 Dec;45(6):401-15. doi: 10.1016/j.ypmed.2007.07.017. Epub 2007 Jul 21. PMID 17707498
- [Background] Fox KR. The influence of physical activity on mental well-being. Public Health Nutr. 1999 Sep;2(3A):411-8. doi: 10.1017/s1368980099000567. PMID 10610081
- [Background] Paluska SA, Schwenk TL. Physical activity and mental health: current concepts. Sports Med. 2000 Mar;29(3):167-80. doi: 10.2165/00007256-200029030-00003. PMID 10739267
- [Background] Bohm AW, Mielke GI, da Cruz MF, Ramirez VV, Wehrmesister FC. Social Support and Leisure-Time Physical Activity Among the Elderly: A Population-Based Study. J Phys Act Health. 2016 Jun;13(6):599-605. doi: 10.1123/jpah.2015-0277. Epub 2015 Dec 21. PMID 26696310
- [Background] Bessey D. Preferences, personality and health behaviors: results from an explorative economic experiment. Int J Health Econ Manag. 2018 Dec;18(4):437-456. doi: 10.1007/s10754-018-9236-1. Epub 2018 Feb 23. PMID 29476285
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Boehm JK, Winning A, Segerstrom S, Kubzansky LD. Variability Modifies Life Satisfaction's Association With Mortality Risk in Older Adults. Psychol Sci. 2015 Jul;26(7):1063-70. doi: 10.1177/0956797615581491. Epub 2015 Jun 5. PMID 26048888
- [Background] Amati V, Meggiolaro S, Rivellini G, Zaccarin S. Social relations and life satisfaction: the role of friends. Genus. 2018;74(1):7. doi: 10.1186/s41118-018-0032-z. Epub 2018 May 4. PMID 29755134
- [Background] Hong SM, Giannakopoulos E. The relationship of satisfaction with life to personality characteristics. J Psychol. 1994 Sep;128(5):547-58. doi: 10.1080/00223980.1994.9914912. PMID 7983611
- [Background] Tugade MM, Fredrickson BL. Resilient individuals use positive emotions to bounce back from negative emotional experiences. J Pers Soc Psychol. 2004 Feb;86(2):320-33. doi: 10.1037/0022-3514.86.2.320. PMID 14769087
- [Background] Hunger C, Bornhauser A, Link L, Geigges J, Voss A, Weinhold J, Schweitzer J. The Experience in Personal Social Systems Questionnaire (EXIS.pers): Development and Psychometric Properties. Fam Process. 2017 Mar;56(1):154-170. doi: 10.1111/famp.12205. Epub 2016 Feb 8. PMID 26858173
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] Koivumaa-Honkanen H, Honkanen R, Viinamaki H, Heikkila K, Kaprio J, Koskenvuo M. Self-reported life satisfaction and 20-year mortality in healthy Finnish adults. Am J Epidemiol. 2000 Nov 15;152(10):983-91. doi: 10.1093/aje/152.10.983. PMID 11092440
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Uchino BN, Uno D, Holt-Lunstad J. Social Support, Physiological Processes, and Health. Curr Dir Psychol Sci. 1999;8(5):145-8
- [Background] Tomasello M, Melis AP, Tennie C, Wyman E, Herrmann E. Two Key Steps in the Evolution of Human Cooperation. Curr Anthropol. [2012;53(6):673-92
- [Background] European Commission. European platform against poverty and social exclusion - A European framework for social and territorial cohesion. 2014. 1-2 p
- [Background] Poverty, social exclusion and health systems in the WHO European Region [Internet]. World Health Organization. 2010 [cited 23 August 2018]. Available from: http://www.euro.who.int/__data/assets/pdf_file/0004/127525/e94499.pdf
- [Background] Jaffee SR, Caspi A, Moffitt TE, Polo-Tomas M, Taylor A. Individual, family, and neighborhood factors distinguish resilient from non-resilient maltreated children: a cumulative stressors model. Child Abuse Negl. 2007 Mar;31(3):231-53. doi: 10.1016/j.chiabu.2006.03.011. Epub 2007 Mar 28. PMID 17395260
- [Background] Gilman R. The Relationship Between Life Satisfaction, Social Interest, and Frequency of Extracurricular Activities Among Adolescent Students. J Youth Adolesc. 2001;30(6):749-67
- [Background] Myers D. Close Relationships and Quality of Life. Well-being: The foundations of hedonic psychology. 1999. 374-391 p.
- [Background] Social Networks, Host Resistance, and Mortality: A Nine-Year Follow-up Study of Alameda County Residents. Am J Epidemiol. 2017 Jun 1;185(11):1070-1088. doi: 10.1093/aje/kwx103. No abstract available. PMID 30052734
- [Background] Waidhofer M. Soziale Kompetenz im Diskurs [Dissertation]. JKU Linz; 2004. German
- [Background] Zautra AJ, Hall JS, Murray KE. Resilience: A New Definition of Health for People and Communities. In: Handbook of Adult Resilience. 2010. p. 3-30
- [Background] Henry JP, Stephens PM. Stress, Health and the Social Environment, A Sociobiologic Approach to Medicine. New York, Heidelberg, Berlin: Springer Verlag; 1977. 282 p.
- [Background] World Health Organization. Promoting Mental Health - Concepts, Emerging Evidence, Practice [Internet]. 2004. Available from: http://www.who.int/mental_health/evidence/en/promoting_mhh.pdf
- [Background] Mental health: a state of well-being [Internet]. World Health Organization. 2014 [cited 26 August 2018]. Available from: http://www.who.int/features/factfiles/mental_health/en/
- [Background] Rhodes RE, Boudreau P. Physical Activity and Personality Traits. Oxford Res Encycl Psychol .2017;1(February):online. Available from: http://psychology.oxfordre.com/view/10.1093/acrefore/9780190236557.001.0001/acrefore-9780190236557-e-210 [Accessed 31 Aug. 2018]
- [Background] Fernández-Ballesteros R, Zamarrón MD, Ruíz MA. The contribution of socio-demographic and psychosocial factors to life satisfaction. Ageing Soc. 2001;21(1):25-43
- [Background] Luhmann M, Lucas RE, Eid M, Diener E. The Prospective Effect of Life Satisfaction on Life Events. Soc Psychol Personal Sci. 2013;4(1):39-45
- [Background] Ryff CD, Singer BH. Know thyself and become what you are: A eudaimonic approach to psychological well-being. J Happiness Stud. 2008;9(1):13-39.
- [Background] Huppert FA. Psychological Well-being: Evidence Regarding its Causes and Consequences. Appl Psychol Heal Well-Being. 2009;1(2):137-64.
- [Background] Reeves BC, Gaus W. Guidelines for reporting non-randomised studies. Forsch Komplementarmed Klass Naturheilkd. 2004 Aug;11 Suppl 1:46-52. doi: 10.1159/000080576. PMID 15353903
- [Background] Kutschera, G. (2018). Entstehung und Entwicklung der Kutschera- Resonanz® Methode. [pdf] Institut Kutschera. Available at: https://www.kutschera.org-/fileadmin/kutschera/pdf/Entwicklung_der_Resonanzmethode.pdf [Accessed 31 Aug. 2018].
- [Background] Tosey P, Langley D, Mathison J. Bateson's Levels Of Learning: a Framework For Workplace Learning. In: van Woerkom M, Poell R, editors. Workplace Learning: Concepts, Measurement, and Application. Routledge; 2010. p. 55-68.
- [Background] Sandu A. Using the Pyramid of Neurological Levels in the Human Resources Motivation Management. Rev Rom pentru Educ Multidimens. 2016;8(2):31-44.
- [Background] Necşoi DV, Porumbu D, Beldianu IF. Self-Reflexivity - Transversal Competence in Teachers' Training. Procedia - Soc Behav Sci. 2013;82:186-91.
- [Background] Kutschera G. Tanz zwischen Bewusst-sein und Unbewusst-sein. Paderborn: Junfermann; 2007. 513 p.
- [Background] Kutschera, G. and Hoffmann, A. (2008). Theorie Sozialkompetenz in der Resonanzmethode®. [pdf] Wien: Institut Kutschera. Available at: https://www.kutschera.org/fileadmin/kutschera/pdf/Publikationen/KutscheraG-KutscheraA_2008_Theorie-Sozialkompetenz-in-der-Resonanzmethode.pdf [Accessed 31 Aug. 2018]
- [Background] Kutschera (2015). Ausbildung zum Kutschera-Resonanz Practitioner. [pdf] Institut Kutschera. Available at: https://www.kundenmeister.com/crm/index.php/-filemanager/getById/1869/22/2_Leitfaden_Practitioner.pdf [Accessed 31 Aug. 2018].
- [Background] Stress - Belastungen besser bewältigen [Internet]. Techniker Krankenkasse; 2017 [cited 31 August 2018]. Available from: https://www.tk.de/resource/blob/2023234/5535b9478a9be8fcabb0a1c6ea7f677e/tk-broschuere--stress--data.pdf
- [Background] Aguilar-Raab C, Mühlhan L, Schweitzer J. EVOS - Evaluation of Social Systems. Kemper CJ, Zenger M, Brähler E, editors. Handbuch Kurzskalen psychologischer Merkmale. Berlin: Medizinisch-Wissenschaftliche Verlagsgesellschaft; 2014. S. 72-75.
- [Background] Klusmann U, Trautwein U, Lüdtke O. Intrinsische und extrinsische Lebensziele: Rehabilität und Validität einer deutschen Fassung des Aspirations Index. Diagnostica. 2005;51(1):40-51.
- [Background] Steger MF, Frazier P, Oishi S, Kaler M. The Meaning in Life Questionnaire: Assessing the Presence of and Search for Meaning in Life. J Couns Psychol. 2006;53(1):80-93.
- [Background] Schumacher J, Wilz G, Gunzelmann T, Brahler E. [The Antonovsky Sense of Coherence Scale. Test statistical evaluation of a representative population sample and construction of a brief scale]. Psychother Psychosom Med Psychol. 2000 Dec;50(12):472-82. doi: 10.1055/s-2000-9207. German. PMID 11199111
- [Background] Ruch W, Martínez-Martí ML, Proyer RT, Harzer C. The Character Strengths Rating Form (CSRF): Development and initial assessment of a 24-item rating scale to assess character strengths. Pers Individ Dif. Elsevier Ltd; 2014;68:53-8.
- [Background] Psychiatric Research Unit - WHO Collaborating Centre in Mental Health. WHO (fünf) - Fragebogen zum Wohlbefinden. Hillerod; 1998
- [Derived] Janka C, Stamm T, Heinze G, Dorner TE. A Training Programme for Developing Social and Personal Resources and Its Effects on the Perceived Stress Level in Adults in Daily Life-Study Protocol for a Prospective Cohort Study. Int J Environ Res Public Health. 2022 Dec 28;20(1):523. doi: 10.3390/ijerph20010523. PMID 36612844

DOCUMENTS (4):
  • Informed Consent Form: Group A - Intervention Group (2019-10-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT04165473/ICF_001.pdf
  • Informed Consent Form: Group B - Intervention Group - Close Relationship (2019-10-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT04165473/ICF_002.pdf
  • Informed Consent Form: Group C - Control Group (2019-10-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT04165473/ICF_003.pdf
  • Informed Consent Form: Group D - Control Group - Close Relationship (2019-10-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT04165473/ICF_004.pdf